CLINICAL TRIAL: NCT02493049
Title: Randomized, Controlled Pilot Trial of Domperidone in Relapsing-Remitting Multiple Sclerosis
Brief Title: Pilot Trial of Domperidone in Relapsing-Remitting Multiple Sclerosis (RRMS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Dr. Luanne Metz, Neurologist, Professor of Clinical Neurosciences, MD, FRCPC, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOM-RRMS-01
Record Dates: First submitted 2015-07-02; First posted 2015-07-09 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Domperidone; Relapsing-Remitting MS; Demyelinating disease; Remyelination
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Demyelinating Diseases | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Domperidone (Experimental): Add on oral Domperidone 10 mg, three times daily. Target dose:30mg daily. Duration: 16 weeks
  Interventions: Drug: Domperidone
- No add on treatment (No Intervention): No add on treatment. Control group

INTERVENTIONS:
Drug: Domperidone — Addition of Domperidone to current Disease Modifying Therapy.
  Other Names: domperidone maleate
  Arms: Domperidone

SUMMARY:
The first major objective of this pilot trial is to demonstrate that it is possible to study myelin repair in relapsing-remitting multiple sclerosis (RRMS) patients with enhancing lesions on MRI by using advanced imaging techniques. To demonstrate that this is possible the investigators will recruit 24 RRMS patients who are being treated with standard disease modifying therapy (DMT) and have new lesions identified on clinically indicated brain MRI scans and measure myelin repair at 16 and 32 weeks using MRI measures of myelin repair. The second major objective is to determine how much repair occurs in participants treated with domperidone compared with those who are not treated. This will allow us to design larger trials to confirm that domperidone improves repair. The study will also confirm the safety and tolerability of domperidone in RRMS, determine circulating prolactin levels during dosing with domperidone 10mg three times daily in people with RRMS, and explore the impact of other clinical factors (such as age) on lesion repair.

In addition, blood will be collected to test for metabolomics and the investigators will bank blood for future study of biomarkers that can help the investigators better understand MS. Metabolomics is an experimental test where changes in the pattern of the chemicals in blood cells are compared at different time points (during and after inflammation). There will be random changes but changes that are common in most study participants may help identify chemicals that signal stages in injury or repair. The investigators will also compare the pattern of change in those with the best repair to those with the worst repair. This may help identify a chemical that is associated with better or worse repair and help develop new treatment strategies. There are currently no blood tests that help in the diagnosis of MS, help determine which drug a person will respond to, or help determine a person's expected MS outcome. Any such tests would be considered biomarkers.

DETAILED DESCRIPTION:
Primary Objectives:

* To demonstrate that the investigators can recruit DMT treated RRMS patients who have breakthrough enhancing lesions identified on clinically indicated monitoring brain MRI scans and measure lesion repair over 32 weeks.
* To obtain estimates of the magnitude and variability of lesion repair in DMT treated RRMS patients who are taking add-on domperidone, or no add-on treatment. The investigators will evaluate three MRI measures [texture analysis, diffusion tensor imaging (DTI), and magnetization transfer imaging (MTI)] for their ability to measure repair within acute enhancing lesions in RRMS. They will also evaluate repair at 16 and 32 weeks. These outcomes will aid in the development of future trials.

No therapies have yet been shown to improve lesion repair, and there is no accepted trial model to evaluate lesion repair in humans. Therefore, the investigators anticipate that the data from this trial will inform the design of future phase 2 trials of therapies to promote lesion repair in MS.

Secondary Objectives:

* To determine the safety and tolerability of domperidone in RRMS
* To determine serum prolactin levels during dosing with domperidone 10mg tid in this population
* To explore metabolomic profiling during lesion repair.
* To explore the impact of the following variables on lesion repair: prolactin level at 6 weeks, concurrent use of each type of DMT, Vitamin D and B12 levels at baseline, patient clinical characteristics (MS duration, EDSS), imaging characteristics (T2 lesion volume, enhancing lesion volume), patient demographics and behaviours (age, sex, smoking status).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between age 18 and 60 years.
* Sexually active men and women of child-bearing potential, defined as those who are not postmenopausal (24 consecutive months) or permanently sterilised, must agree to use adequate contraception. Adequate contraception is defined as methods of birth control which result in a low failure rate [i.e. less than 1% per year] when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), barrier contraceptives, sexual abstinence or vasectomised partner. Adequate contraception is required during domperidone treatment and for one month after stopping treatment.
* Participants must have MS defined according to the McDonald criteria (Polman et al. 2011).
* Participants must have RRMS according to Lublin et al. (2014).
* Participants must have been treated with a stable approved dose of glatiramer acetate, interferon-beta, fingolimod, dimethyl fumarate, or teriflunomide for at least 6 months.
* Participants must be scheduled to have a clinically indicated brain MRI to monitor DMT effectiveness.
* Participants must have at least one gadolinium enhancing lesion on their DMT monitoring MRI (screening MRI).
* Participants must report at least 80% adherence to their current DMT and have had no treatment discontinuation for one week or longer within the prior 6 months.
* Participants must be patients of the Calgary MS Clinic.
* Participants must provide written informed consent

Exclusion Criteria:

* Participants who are pregnant or breastfeeding
* Participants in whom it is expected that their current DMT will be discontinued within 16 weeks. Indicators of likely discontinuation will include poor DMT tolerance, a wish by the participant to discontinue the DMT, or a history of poor clinical response to the current DMT (such as a relapse within the previous year while on the current DMT)
* Participants who have a long QT interval, defined as corrected QT interval of more than 470 msec in men and more than 450 msec in women, on screening ECG.
* Participants with known long-QT syndrome or known cardiac arrhythmia.
* Participants who currently or previously have been treated with natalizumab.
* Participants who are currently treated with domperidone or have taken it within the previous 3 months.
* Participants who are taking drugs which prolong QT intervals or who are treated with drugs that inhibit cytochrome P450 3A4.
* Participants who are concurrently treated with drugs that may increase serum prolactin levels.
* Participants who have a prolactinoma
* Participants who use systemic corticosteroids within the 8 weeks prior to the screening MRI or who use concurrent immunosuppressive medications including systemic corticosteroids.
* Participants who have a history of breast cancer or breast carcinoma in situ or who have clinically significant depression, renal, hepatic, cardiovascular, respiratory, metabolic, ophthalmologic, cerebrovascular, or other serious physical disease.
* Participants in whom gastrointestinal stimulation might be dangerous, i.e. gastrointestinal hemorrhage or mechanical obstruction or perforation
* Participants who have a known allergy or other intolerability to domperidone.
* Participants with serum potassium, sodium, magnesium or calcium levels outside the normal range, serum creatinine > 6 mg/100 ml or > 0.6 mmol/l), or who have any other condition or situation that in the opinion of the investigator would either put the patient at risk of worsening health if enrolled in the trial or would prevent completion of the trial.
* Participants who are concurrently participating in any therapeutic clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Measures of repair within enhancing T1 MRI lesions | up to 32 weeks
  Texture analysis, Diffusion Tensor Imaging (DTI) and Magnetization Transfer Imaging (MTI) will be used. This is a pilot study so the investigators are measuring repair at 2 time points and with 3 imaging methods to aid in the design of future studies.

SECONDARY OUTCOMES:
Number and type of adverse events over the 16 week treatment period. | at 6 and 16 weeks
  Adverse events will be collected at all visits and by telephone if an encounter occurs. Clinical outcomes are not sufficiently sensitive or specific to stand as measures of repair in phase 2 clinical trials that aim to screen therapies for their potential to provide neuroprotection or enhance repair. Therefore the investigators will only use clinical measures at the baseline visit to describe participants with regards to level of clinical impairment. The investigators will use the standard measure of clinical impairment, the EDSS. The baseline neurological examination and EDSS will also be used to confirm the occurrence of a relapse. A relapse that occurs during the treatment period in a participant on domperidone will be considered an adverse event. Enhancing lesions on MRI after baseline will also be considered adverse events.
Serum Prolactin Levels at both 6 and 16 weeks | at 6 and 16 weeks
  To determine how much domperidone 10mg three times daily increases serum prolactin levels in this MS population over time. The investigators will also explore the relationship between prolactin level and repair.

CONTACTS AND LOCATIONS:
Overall Officials: Luanne M Metz, MD, Principal Investigator — University of Calgary
Locations (1):
- Calgary MS Clinic at Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
consent to share IPD was not obtained so we cannot share

REFERENCES:
- [Background] Alonso-Ortiz E, Levesque IR, Pike GB. MRI-based myelin water imaging: A technical review. Magn Reson Med. 2015 Jan;73(1):70-81. doi: 10.1002/mrm.25198. Epub 2014 Mar 6. PMID 24604728
- [Background] Bagnato F, Jeffries N, Richert ND, Stone RD, Ohayon JM, McFarland HF, Frank JA. Evolution of T1 black holes in patients with multiple sclerosis imaged monthly for 4 years. Brain. 2003 Aug;126(Pt 8):1782-9. doi: 10.1093/brain/awg182. Epub 2003 Jun 23. PMID 12821527
- [Background] Barkhof F, Bruck W, De Groot CJ, Bergers E, Hulshof S, Geurts J, Polman CH, van der Valk P. Remyelinated lesions in multiple sclerosis: magnetic resonance image appearance. Arch Neurol. 2003 Aug;60(8):1073-81. doi: 10.1001/archneur.60.8.1073. PMID 12925362
- [Background] Barkhof F, Calabresi PA, Miller DH, Reingold SC. Imaging outcomes for neuroprotection and repair in multiple sclerosis trials. Nat Rev Neurol. 2009 May;5(5):256-66. doi: 10.1038/nrneurol.2009.41. PMID 19488083
- [Background] Bernini GP, Lucarini AR, Franchi F, Salvetti A. Humoral effects of metoclopramide and domperidone in normal subjects and in hypertensive patients. J Endocrinol Invest. 1988 Nov;11(10):711-6. doi: 10.1007/BF03350925. PMID 2852692
- [Background] Lublin FD, Baier M, Cutter G. Effect of relapses on development of residual deficit in multiple sclerosis. Neurology. 2003 Dec 9;61(11):1528-32. doi: 10.1212/01.wnl.0000096175.39831.21. PMID 14663037
- [Background] Filippi M, Rovaris M, Rocca MA, Sormani MP, Wolinsky JS, Comi G; Eurpoean/Canadian Glatiramer Acetate Study Group. Glatiramer acetate reduces the proportion of new MS lesions evolving into "black holes". Neurology. 2001 Aug 28;57(4):731-3. doi: 10.1212/wnl.57.4.731. PMID 11524494
- [Background] Trapp BD, Peterson J, Ransohoff RM, Rudick R, Mork S, Bo L. Axonal transection in the lesions of multiple sclerosis. N Engl J Med. 1998 Jan 29;338(5):278-85. doi: 10.1056/NEJM199801293380502. PMID 9445407
- [Background] Bjartmar C, Kidd G, Mork S, Rudick R, Trapp BD. Neurological disability correlates with spinal cord axonal loss and reduced N-acetyl aspartate in chronic multiple sclerosis patients. Ann Neurol. 2000 Dec;48(6):893-901. PMID 11117546
- [Background] Metz LM, Zhang Y, Yeung M, Patry DG, Bell RB, Stoian CA, Yong VW, Patten SB, Duquette P, Antel JP, Mitchell JR. Minocycline reduces gadolinium-enhancing magnetic resonance imaging lesions in multiple sclerosis. Ann Neurol. 2004 May;55(5):756. doi: 10.1002/ana.20111. No abstract available. PMID 15122721
- [Background] Sloka S, Metz LM, Hader W, Starreveld Y, Yong VW. Reduction of microglial activity in a model of multiple sclerosis by dipyridamole. J Neuroinflammation. 2013 Jul 18;10:89. doi: 10.1186/1742-2094-10-89. PMID 23866809
- [Background] Chandran S, Hunt D, Joannides A, Zhao C, Compston A, Franklin RJ. Myelin repair: the role of stem and precursor cells in multiple sclerosis. Philos Trans R Soc Lond B Biol Sci. 2008 Jan 12;363(1489):171-83. doi: 10.1098/rstb.2006.2019. PMID 17282989
- [Background] Franklin RJ. Why does remyelination fail in multiple sclerosis? Nat Rev Neurosci. 2002 Sep;3(9):705-14. doi: 10.1038/nrn917. PMID 12209119
- [Background] Zhao C, Fancy SP, Kotter MR, Li WW, Franklin RJ. Mechanisms of CNS remyelination--the key to therapeutic advances. J Neurol Sci. 2005 Jun 15;233(1-2):87-91. doi: 10.1016/j.jns.2005.03.008. PMID 15949498
- [Background] Gregg C, Shikar V, Larsen P, Mak G, Chojnacki A, Yong VW, Weiss S. White matter plasticity and enhanced remyelination in the maternal CNS. J Neurosci. 2007 Feb 21;27(8):1812-23. doi: 10.1523/JNEUROSCI.4441-06.2007. PMID 17314279
- [Background] Xiao L, Xu H, Zhang Y, Wei Z, He J, Jiang W, Li X, Dyck LE, Devon RM, Deng Y, Li XM. Quetiapine facilitates oligodendrocyte development and prevents mice from myelin breakdown and behavioral changes. Mol Psychiatry. 2008 Jul;13(7):697-708. doi: 10.1038/sj.mp.4002064. Epub 2007 Aug 7. PMID 17684494
- [Background] Mi S, Pepinsky RB, Cadavid D. Blocking LINGO-1 as a therapy to promote CNS repair: from concept to the clinic. CNS Drugs. 2013 Jul;27(7):493-503. doi: 10.1007/s40263-013-0068-8. PMID 23681979
- [Background] Nerozzi D, Magnani A, Dastoli C, Ferri E, Capesciotti G, Antonozzi I, Frajese G, Meltzer HY. Prolactin responses to domperidone in chronic schizophrenia. Psychiatry Res. 1992 May;42(2):159-69. doi: 10.1016/0165-1781(92)90079-i. PMID 1631251
- [Background] Knoppert DC, Page A, Warren J, Seabrook JA, Carr M, Angelini M, Killick D, Dasilva OP. The effect of two different domperidone doses on maternal milk production. J Hum Lact. 2013 Feb;29(1):38-44. doi: 10.1177/0890334412438961. Epub 2012 May 3. PMID 22554679
- [Background] Mallik S, Samson RS, Wheeler-Kingshott CA, Miller DH. Imaging outcomes for trials of remyelination in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2014 Dec;85(12):1396-404. doi: 10.1136/jnnp-2014-307650. Epub 2014 Apr 25. PMID 24769473
- [Derived] Zhang Y, Liu WQ, Hosseinpour Z, Pike GB, Cerchiaro G, Greenfield J, Yong VW, Metz LM. Feasibility study to assess lesion repair in relapsing-remitting multiple sclerosis: A randomized controlled pilot clinical trial of domperidone add-on treatment. Mult Scler Relat Disord. 2024 May;85:105525. doi: 10.1016/j.msard.2024.105525. Epub 2024 Feb 27. PMID 38461731